CLINICAL TRIAL: NCT00006036
Title: A Phase I Study of NX 211 in Combination With Cisplatin Given as an IV Infusion Days 1, 2, and 3 Every 3 Weeks in Patients With Solid Tumors
Brief Title: Liposomal Lurtotecan Plus Cisplatin in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I133; CAN-NCIC-IND133 (Other: PDQ); NEXSTAR-110-05 (Other: Nexstar); CDR0000068051 (Other: PDQ)
Record Dates: First submitted 2000-07-05; First posted 2004-03-25 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Cancer; Lung Cancer; Ovarian Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent non-small cell lung cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage IV nasopharyngeal cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; ovarian stromal cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Nasopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: lurtotecan liposome

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of liposomal lurtotecan plus cisplatin in treating patients who have advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and recommended phase II dose of lurtotecan liposome and cisplatin in patients with advanced solid tumors. II. Determine the toxicity profile, dose-limiting toxic effects, and the pharmacokinetics of this treatment regimen in this patient population. III. Determine any correlation between toxicity profile and pharmacokinetics of this treatment regimen in these patients. IV. Determine the objective tumor response to this treatment regimen in patients with measurable disease (previously untreated solid tumors) entered at the recommended phase II dose.

OUTLINE: This is an open-label, multicenter, dose-escalation study of lurtotecan liposome. Patients receive cisplatin IV over 1 hour followed by lurtotecan liposome IV over 30 minutes on days 1-3. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Once the total dose of cisplatin is reached, patients receive lurtotecan liposome alone. Patients achieving complete response (CR) continue therapy for 2 courses after documentation of confirmed CR. Patients achieving partial response (PR) continue therapy until progression or for 2 courses after documentation of stable PR. Patients with stable disease continue therapy for a maximum of 6 courses. Cohorts of 3-6 patients receive escalating doses of lurtotecan liposome until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 10 patients with previously untreated solid tumors are treated at the recommended phase II dose (1 dose below the MTD). Patients are followed at 4 weeks and then every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 20-25 patients will be accrued for this study within 12-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced and/or metastatic solid tumor refractory to standard curative therapy or for which no curative therapy exists Clinically or radiographically documented disease No tumor marker elevation as only evidence of disease No untreated brain or meningeal metastases Previously treated and stable CNS metastases allowed (i.e., no evidence of increasing disease by CT scan for at least 4 weeks) Recommended phase II dose portion of study: Previously untreated advanced and/or metastatic disease for which a cisplatin-based regimen is indicated (e.g., non-small cell lung cancer, small cell lung cancer, ovarian, or head and neck cancer) At least one measurable lesion at least 20 mm by physical exam or x-ray or at least 10 mm by spiral CT scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST/ALT no greater than 2.5 times ULN (5 times ULN if documented liver metastases) Renal: Creatinine no greater than ULN OR Creatinine clearance at least 60 mL/min Other: No greater than grade 1 neuropathy or ototoxicity No other prior or concurrent malignancy within the past 5 years except curatively treated basal or squamous cell skin cancer or cervical cancer (for recommended phase II dose) No active or uncontrolled infections No other serious illnesses or medical conditions that would preclude study No known hypersensitivity to systemic liposomal formulation or any drug chemically related to study drug Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Chemotherapy Recovered from prior immunotherapy Chemotherapy: See Disease Characteristics No more than 1 prior chemotherapy regimen (adjuvant and/or metastatic) except for nonmyelosuppressive agents (e.g., signal transduction inhibitors or immunotherapy) At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin and 4 weeks for carboplatin) and recovered At least 1 year since prior high-dose chemotherapy with marrow or stem cell support No prior total cisplatin dose of more than 300 mg/m2 No prior chemotherapy (for recommended phase II dose) Endocrine therapy: Prior hormonal therapy allowed Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior radiotherapy to more than 25% of bone marrow reserve, except for low-dose nonmyelosuppression Surgery: Not specified Other: At least 4 weeks since other prior experimental drugs or anticancer therapy and recovered No other concurrent investigational or anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2000-03-22 (Actual); Primary Completion 2002-09-26 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hal W. Hirte, MD, FRCP(C), Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (3):
- Canada (3):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MacKenzie MJ, Hirte HW, Siu LL, Gelmon K, Ptaszynski M, Fisher B, Eisenhauer E. A phase I study of OSI-211 and cisplatin as intravenous infusions given on days 1, 2 and 3 every 3 weeks in patients with solid cancers. Ann Oncol. 2004 Apr;15(4):665-70. doi: 10.1093/annonc/mdh133. PMID 15033677